CLINICAL TRIAL: NCT00389207
Title: Randomized, Open Label Study Evaluating the Lipid Profile Difference and Efficacy of a Combined Therapy Including Tenofovir, Emtricitabine + Atazanavir / r or NVP in Naive HIV - 1 Infected Patients.
Brief Title: Nevirapine or Atazanavir/Ritonavir Given With Emtricitabine/Tenofovir in Human Immunodeficiency Virus (HIV)-1-infected Treatment Naive Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1100.1470; 2005-004330-40 (EudraCT Number: EudraCT)
Record Dates: First submitted 2006-10-17; First posted 2006-10-18 (Estimated); Results first posted 2012-03-26 (Estimated); Last update posted 2014-01-27 (Estimated); Status verified 2013-12

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Atazanavir Sulfate

ARMS (3):
- NVP bid (Active Comparator): nevirapine (NVP) 200 mg BID in combination with emtricitabine (FTC) and tenofovir DF (TDF)
  Interventions: Drug: nevirapine bid
- NVP qd (Experimental): nevirapine (NVP) 400 mg QD in combination with emtricitabine (FTC) and tenofovir DF (TDF)
  Interventions: Drug: nevirapine qd
- ATZ/r (Active Comparator): ritonavir-boosted atazanavir in combination with emtricitabine (FTC) and tenofovir DF (TDF)
  Interventions: Drug: atazanavir

INTERVENTIONS:
Drug: nevirapine bid — nevirapine twice daily
  Arms: NVP bid
Drug: nevirapine qd — nevirapine once daily
  Arms: NVP qd
Drug: atazanavir — atazanavir once daily
  Arms: ATZ/r

SUMMARY:
Primary purpose of this study is to compare the efficacy and safety of two different nevirapine (Viramune) dosing regimens (once daily (QD) and twice daily (BID) application) and of atazanavir/ritonavir (Reyataz/Norvir), all on an emtricitabine/tenofovir disoproxil fumarate (DF) (Truvada) background. Patients will receive either nevirapine (NVP) 200 mg twice daily, or NVP 400 mg once daily , or ritonavir-boosted atazanavir (ATZ/r), all in combination with emtricitabine (FTC) and tenofovir DF (TDF).

All patients receiving NVP will start at 200 mg once daily for 2 weeks, because it has been demonstrated that this lead-in dosing regimen reduces the frequency of NVP-induced rash. At Visit 3 (Week 2), patients increase the NVP dose to either 200 mg twice daily or to 400 mg once daily. Patients receiving ATZ/r will be treated with ATZ 300 mg once daily, boosted by 100 mg ritonavir (RTV) once daily. Background antiretroviral therapy for all patients consists of one tablet of Truvada. Treatment duration is 48 weeks (primary endpoint) with an extension to 144 weeks. Patients may also participate in the metabolic sub-study, comparing NVP and ATZ/r for signs and symptoms of lipodystrophy and serum lipid/glycaemic abnormalities.

ELIGIBILITY:
Inclusion criteria:

Inclusion Criteria:

1. Signed informed consent in accordance with Good Clinical Practice (GCP) and local regulatory requirements prior to trial participation
2. HIV-1-infected males or females >= 18 years of age with positive serology confirmed by Western blot
3. No previous antiretroviral treatment (of more than 7 days)
4. Males with CD4+ counts of < 400 cells/mm3 and females with CD4+ counts of < 250 cells/mm3
5. NVP- and ATZ/r susceptibility based on HIV-1 genotypic resistance report
6. Adequate renal function defined as a calculated creatinine clearance (CLCr) >= 50 ml/min according to the Cockcroft-Gault formula
7. Karnofsky score >= 70
8. Acceptable medical history, as assessed by the investigator

Exclusion criteria:

Exclusion Criteria:

1. Active drug abuse or chronic alcoholism at the investigator's discretion
2. Hepatic cirrhosis stage Child-Pugh B or C
3. Female patients of child-bearing potential who:

   * have a positive serum pregnancy test at screening or during the study,
   * are breast feeding,
   * are planning to become pregnant,
   * are not willing to use a barrier method of contraception, or are not willing to use methods of contraception other than ethinyl estradiol containing oral contraceptives
4. Laboratory parameters Division of Acquired Immunodeficiency Syndrome (DAIDS) > grade 2 (triglycerides > DAIDS grade 3; total cholesterol no restrictions)
5. Active hepatitis B or C disease, defined as HBsAg-positive or Hepatitis C-Virus-Ribo Nucleic Acid (HCV-RNA)- positive with Aspartate Transaminase/Alanine Transaminase (AST/ALT) > 2.5x Upper Limit of Normal (ULN) (DAIDS grade 1)
6. Hypersensitivity to any ingredients of the test products
7. Have therapy with nephrotoxic drugs (e.g., aminoglycosides, amphotericin B, vancomycin, cidofovir, foscarnet, cisplatin, pentamidine, tacrolimus, cyclosporine) or potential competitors of renal excretion (e.g., cidofovir, acyclovir, valacyclovir, ganciclovir, valganciclovir, probenecid, high-dose non-steroidal anti-inflammatory drugs (i.e., ibuprofen)) within 3 months prior to study screening or are expected to receive these during the study
8. Patients who are receiving other concomitant treatments which are not permitted
9. Use of other investigational medications within 30 days before study entry or during the trial
10. Use of immunomodulatory drugs within 30 days before study entry or during the trial (e.g., interferon, cyclosporin, hydroxyurea, interleukin 2, chronic treatment with prednisone)
11. Patients with Progressive Multifocal Leukoencephalopathy (PML), Visceral Kaposi's Sarcoma (KS), and/or any lymphoma
12. Any AIDS defining illness that is unresolved, symptomatic or not stable on treatment for at least 12 weeks at screening visit
13. Patients who are receiving systemic treatment for malignant disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 576 (Actual)
Dates: Start 2006-10; Primary Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (68):
- Argentina (4):
  - 1100.1470.54004 Boehringer Ingelheim Investigational Site, Capital Federal
  - 1100.1470.54002 Boehringer Ingelheim Investigational Site, Córdoba
  - 1100.1470.54003 Boehringer Ingelheim Investigational Site, Mar del Plata
  - 1100.1470.54001 Boehringer Ingelheim Investigational Site, Rosario
- Germany (17):
  - 1100.1470.49001 Boehringer Ingelheim Investigational Site, Berlin
  - 1100.1470.49002 Boehringer Ingelheim Investigational Site, Berlin
  - 1100.1470.49003 Boehringer Ingelheim Investigational Site, Bochum
  - 1100.1470.49018 Boehringer Ingelheim Investigational Site, Bonn
  - 1100.1470.49014 Boehringer Ingelheim Investigational Site, Düsseldorf
  - 1100.1470.49008 Boehringer Ingelheim Investigational Site, Erlangen
  - 1100.1470.49035 Boehringer Ingelheim Investigational Site, Frankfurt
  - 1100.1470.49036 Boehringer Ingelheim Investigational Site, Frankfurt am Main
  - 1100.1470.49033 Boehringer Ingelheim Investigational Site, Freiburg/Breisgau
  - 1100.1470.49016 Boehringer Ingelheim Investigational Site, Hamburg
  - 1100.1470.49031 Boehringer Ingelheim Investigational Site, Hamburg
  - 1100.1470.49037 Boehringer Ingelheim Investigational Site, Hamburg
  - 1100.1470.49020 Boehringer Ingelheim Investigational Site, Hanover
  - 1100.1470.49038 Boehringer Ingelheim Investigational Site, Magdeburg
  - 1100.1470.49034 Boehringer Ingelheim Investigational Site, München
  - 1100.1470.49000 Boehringer Ingelheim Investigational Site, Ulm
  - 1100.1470.49032 Boehringer Ingelheim Investigational Site, Würzburg
- Italy (8):
  - 1100.1470.39001 Boehringer Ingelheim Investigational Site, Bergamo
  - 1100.1470.39003 Boehringer Ingelheim Investigational Site, Bologna
  - 1100.1470.39012 Ospedale Sant'Anna, Como
  - 1100.1470.39006 Boehringer Ingelheim Investigational Site, Ferrara
  - 1100.1470.39010 Boehringer Ingelheim Investigational Site, Lecco
  - 1100.1470.39004 Boehringer Ingelheim Investigational Site, Torino
  - 1100.1470.39009 Boehringer Ingelheim Investigational Site, Torrette Di Ancona
  - 1100.1470.39007 Boehringer Ingelheim Investigational Site, Varese
- Mexico (6):
  - 1100.1470.55006 Boehringer Ingelheim Investigational Site, Aguascalientes
  - 1100.1470.55004 Boehringer Ingelheim Investigational Site, Col Obregón
  - 1100.1470.55008 Boehringer Ingelheim Investigational Site, Col. Los Filtros, San Luis Potosí
  - 1100.1470.55001 Boehringer Ingelheim Investigational Site, Col. Toriello Guerra
  - 1100.1470.55007 Boehringer Ingelheim Investigational Site, Guadalajara Jal.
  - 1100.1470.55003 Boehringer Ingelheim Investigational Site, Tlalpan-México D,F
- Poland (4):
  - 1100.1470.48003 Boehringer Ingelheim Investigational Site, Bydgoszcz
  - 1100.1470.48001 Boehringer Ingelheim Investigational Site, Chorzów
  - 1100.1470.48002 Boehringer Ingelheim Investigational Site, Szczecin
  - 1100.1470.48004 Boehringer Ingelheim Investigational Site, Warsaw
- Portugal (3):
  - 1100.1470.35102 Boehringer Ingelheim Investigational Site, Cascais
  - 1100.1470.35101 Boehringer Ingelheim Investigational Site, Lisbon
  - 1100.1470.35103 Boehringer Ingelheim Investigational Site, Porto
- Romania (2):
  - 1100.1470.40001 Boehringer Ingelheim Investigational Site, Bucharest
  - 1100.1470.40002 Boehringer Ingelheim Investigational Site, Bucharest
- Spain (14):
  - 1100.1470.34013 Boehringer Ingelheim Investigational Site, Alcalá de Henares (Madrid)
  - 1100.1470.34008 Boehringer Ingelheim Investigational Site, Badalona
  - 1100.1470.34002 Boehringer Ingelheim Investigational Site, Barcelona
  - 1100.1470.34003 Boehringer Ingelheim Investigational Site, Barcelona
  - 1100.1470.34004 Boehringer Ingelheim Investigational Site, Donostia / San Sebastian
  - 1100.1470.34009 Boehringer Ingelheim Investigational Site, L'Hospitalet de Llobregat
  - 1100.1470.34010 Boehringer Ingelheim Investigational Site, Madrid
  - 1100.1470.34012 Boehringer Ingelheim Investigational Site, Madrid
  - 1100.1470.34014 Boehringer Ingelheim Investigational Site, Madrid
  - 1100.1470.34015 Boehringer Ingelheim Investigational Site, Madrid
  - 1100.1470.34019 Boehringer Ingelheim Investigational Site, Málaga
  - 1100.1470.34007 Boehringer Ingelheim Investigational Site, Sabadell (Barcelona)
  - 1100.1470.34006 Boehringer Ingelheim Investigational Site, Santa Cruz de Tenerife
  - 1100.1470.34011 Boehringer Ingelheim Investigational Site, Vigo
- Switzerland (4):
  - 1100.1470.41004 Boehringer Ingelheim Investigational Site, Bern
  - 1100.1470.41001 Boehringer Ingelheim Investigational Site, Lugano
  - 1100.1470.41003 Boehringer Ingelheim Investigational Site, Sankt Gallen
  - 1100.1470.41002 Boehringer Ingelheim Investigational Site, Zurich
- United Kingdom (6):
  - 1100.1470.44004 Boehringer Ingelheim Investigational Site, Birmingham
  - 1100.1470.44001 Boehringer Ingelheim Investigational Site, London
  - 1100.1470.44002 Boehringer Ingelheim Investigational Site, London
  - 1100.1470.44005 Boehringer Ingelheim Investigational Site, London
  - 1100.1470.44006 Boehringer Ingelheim Investigational Site, London
  - 1100.1470.44003 Boehringer Ingelheim Investigational Site, Manchester

REFERENCES:
- [Derived] Seclen E, Soriano V, Gonzalez MM, Martin-Carbonero L, Gellermann H, Distel M, Kadus W, Poveda E. Impact of baseline HIV-1 tropism on viral response and CD4 cell count gains in HIV-infected patients receiving first-line antiretroviral therapy. J Infect Dis. 2011 Jul 1;204(1):139-44. doi: 10.1093/infdis/jir218. PMID 21628668
- [Derived] Soriano V, Arasteh K, Migrone H, Lutz T, Opravil M, Andrade-Villanueva J, Antunes F, Di Perri G, Podzamczer D, Taylor S, Domingo P, Gellermann H, de Rossi L; ARTEN investigators. Nevirapine versus atazanavir/ritonavir, each combined with tenofovir disoproxil fumarate/emtricitabine, in antiretroviral-naive HIV-1 patients: the ARTEN Trial. Antivir Ther. 2011;16(3):339-48. doi: 10.3851/IMP1745. PMID 21555816

RESULTS

PARTICIPANT FLOW:
Groups:
- Nevirapine QD: Nevirapine (NVP) 400mg QD on a background of the fixed combination Truvada® (emitricitabine 200mg QD and tenofovir 300mg QD)
- Nevirapine BID: NVP 200mg BID on a background of the fixed combination Truvada®
- Atazanvir/Ritonavir: Atazanvir 300mg QD boosted by ritonavir 100mg QD (ATZ/r) on a background of the fixed combination Truvada®
Period: Overall Study
Arm/Group | Nevirapine QD | Nevirapine BID | Atazanvir/Ritonavir
Started | 188 (3 patients were randomized to NVP QD but not treated and so not part of the Full Analysis Set (FAS)) | 188 (4 patients were randomized to NVP BID but not treated and so are not part of the FAS) | 193
Completed | 125 | 116 | 152
Not Completed | 63 | 72 | 41
Not completed — Adverse Event | 26 | 32 | 10
Not completed — Protocol Violation | 3 | 1 | 4
Not completed — Lost to Follow-up | 12 | 9 | 7
Not completed — Withdrawal by Subject | 5 | 7 | 11
Not completed — Other | 17 | 23 | 9

BASELINE CHARACTERISTICS:
Groups:
- Atazanvir/Ritonavir: ATZ/r on a background of the fixed combination Truvada®
- Total: Total of all reporting groups
Arm/Group | Nevirapine QD | Nevirapine BID | Atazanvir/Ritonavir | Total
Number analyzed (Participants) | 188 | 188 | 193 | 569
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.4 (9.7) | 40.0 (10.5) | 37.6 (9.5) | 38.6 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 25 | 31 | 92
  Male | 152 | 163 | 162 | 477
Baseline HIV viral load category [Number; unit: participants]
  Baseline HIV viral load ≤ 100,000 copies/mL | 71 | 71 | 65 | 207
  Baseline HIV viral load > 100,000 copies/mL | 117 | 117 | 128 | 362
Baseline log10 HIV viral load [Mean (Standard Deviation); unit: log 10 Copies/mL] — 185 NVP QD patients, 188 NVP BID patients and 192 ATZ/R patients had data
  log 10 Copies/mL | 5.1 (0.7) | 5.1 (0.6) | 5.1 (0.7) | 5.1 (0.7)
Baseline CD4+ cell count [Mean (Standard Deviation); unit: Cells/mm^3] — 185 NVP QD patients, 188 NVP BID patients and 192 ATZ/R patients had data
  Cells/mm^3 | 183.3 (95.5) | 202.9 (93.6) | 193.2 (95.8) | 193.2 (95.1)

OUTCOME MEASURES:

1. Primary Outcome: Treatment Response at Week 48
Description: Treatment response is defined as a viral load (VL) <50 copies/mL measured at two consecutive visits prior to Week 48 and without subsequent rebound or change of antiretroviral (ARV) therapy prior to Week 48.
Time Frame: From baseline to Week 48
Population: Full Analysis Set (FAS) defined as all randomized and treated patients but numbers are reduced as indicated due to empty cells in analyses adjusting for baseline categories
Measure: Number; unit: Patients
Groups:
- Nevirapine QD+BID: NVP 400mg QD or 200mg BID on a background of the fixed combination Truvada®
Arm/Group | Nevirapine QD | Nevirapine BID | Nevirapine QD+BID | Atazanvir/Ritonavir
Number analyzed (Participants) | 188 | 188 | 376 | 193
Patients
  Number of responders | 126 | 124 | 250 | 126
  Number of non-responders | 62 | 64 | 126 | 67
Statistical Analysis 1: Comparison: Nevirapine QD+BID vs Atazanvir/Ritonavir; Test type: Non-Inferiority or Equivalence — Non-inferiority margin 12% (or 0.12 as proportion); p = 0.684, Cochran-Mantel-Haenszel — Test for superiority following confirmation of non-inferiority; Controlling for screening VL and CD4+ categories (only 373 NVP patients due to empty cells); Risk Difference (RD) = 0.016, 95% CI [-0.062 to 0.095]
Statistical Analysis 2: Comparison: Nevirapine QD vs Atazanvir/Ritonavir; Test type: Non-Inferiority or Equivalence — Non-inferiority margin 12% (or 0.12 as proportion); p = 0.584, Cochran-Mantel-Haenszel — Test for superiority following confirmation of non-inferiority; Analysis controlling for screening viral load and CD4+ count categories. N=186 NVP QD patients and N=193 ATZ/r patients; Risk Difference (RD) = 0.025, 95% CI [-0.065 to 0.115]
Statistical Analysis 3: Comparison: Nevirapine BID vs Atazanvir/Ritonavir; Test type: Non-Inferiority or Equivalence — Non-inferiority margin 12% (or 0.12 as proportion); p = 0.855, Cochran-Mantel-Haenszel — Test for superiority following confirmation of non-inferiority; Analysis controlling for screening viral load and CD4+ count categories. N=187 NVP QD patients and N=193 ATZ/r patients; Risk Difference (RD) = 0.009, 95% CI [-0.084 to 0.101]

2. Secondary Outcome: Treatment Response at Week 48 (TLOVR Algorithm)
Description: Treatment response is defined as a VL <50 copies/mL measured at two consecutive visits up to Week 48 and without subsequent rebound or change of ARV therapy up to Week 48, based on time to loss of virologic response (TLOVR) algorithm, as a sensitivity analysis for the primary analysis.
Time Frame: From baseline to Week 48
Population: FAS but numbers are reduced as indicated due to empty cells in analysis adjusting for baseline categories
Measure: Number; unit: Patients
Arm/Group | Nevirapine QD+BID | Atazanvir/Ritonavir
Number analyzed (Participants) | 376 | 193
Patients
  Number of responders | 261 | 142
  Number of non-responders | 115 | 51
Statistical Analysis 1: Comparison: Nevirapine QD+BID vs Atazanvir/Ritonavir; Test type: Non-Inferiority or Equivalence — Non-inferiority margin 12% (or 0.12 as proportion); p = 0.321, Cochran-Mantel-Haenszel — Test for superiority following confirmation of non-inferiority; Analysis controlling for screening viral load and CD4+ count categories. N=373 NVP QD patients and N=193 ATZ/r patients; Risk Difference (RD) = -0.038, 95% CI [-0.112 to 0.037]

3. Secondary Outcome: Proportion of Patients With VL < 50 Copies/ml
Description: VL <50 copies/mL among observed patients on treatment at each visit, with the final visit at Week 144 or end of trial (EOT) for the patient
Time Frame: From baseline to Weeks 4, 8, 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, 132 and 144/EOT
Population: FAS with varying numbers missing or not on treatment per visit
Measure: Number; unit: Proportion of patients
Arm/Group | Nevirapine QD+BID | Atazanvir/Ritonavir
Number analyzed (Participants) | 376 | 193
Proportion of patients
  Proportion with VL<50 copies /mL at Week 4 | 0.107 | 0.09
  Proportion with VL<50 copies /mL at Week 8 | 0.304 | 0.25
  Proportion with VL<50 copies /mL at Week 12 | 0.515 | 0.412
  Proportion with VL<50 copies /mL at Week 24 | 0.842 | 0.779
  Proportion with VL<50 copies /mL at Week 36 | 0.907 | 0.83
  Proportion with VL<50 copies /mL at Week 48 | 0.931 | 0.886
  Proportion with VL<50 copies /mL at Week 60 | 0.959 | 0.901
  Proportion with VL<50 copies /mL at Week 72 | 0.965 | 0.915
  Proportion with VL<50 copies /mL at Week 84 | 0.972 | 0.896
  Proportion with VL<50 copies /mL at Week 96 | 0.98 | 0.924
  Proportion with VL<50 copies /mL at Week 108 | 0.964 | 0.968
  Proportion with VL<50 copies /mL at Week 120 | 0.976 | 0.955
  Proportion with VL<50 copies /mL at Week 132 | 0.971 | 0.947
  Proportion with VL<50 copies /mL at Week 144/EOT | 0.952 | 0.929

4. Secondary Outcome: Proportion of Patients With VL < 400 Copies/ml
Description: VL <400 copies/mL among observed patients on treatment at each visit, with the final visit at Week 144 or end of trial (EOT)
Time Frame: From baseline to Weeks 4, 8, 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, 132 and 144/EOT
Population: FAS with varying numbers missing or not on treatment per visit
Measure: Number; unit: Proportion of patients
Arm/Group | Nevirapine QD+BID | Atazanvir/Ritonavir
Number analyzed (Participants) | 376 | 193
Proportion of patients
  Proportion with VL<400 copies /mL at Week 4 | 0.365 | 0.287
  Proportion with VL<400 copies /mL at Week 8 | 0.714 | 0.679
  Proportion with VL<400 copies /mL at Week 12 | 0.856 | 0.834
  Proportion with VL<400 copies /mL at Week 24 | 0.924 | 0.956
  Proportion with VL<400 copies /mL at Week 36 | 0.968 | 0.966
  Proportion with VL<400 copies /mL at Week 48 | 0.985 | 0.977
  Proportion with VL<400 copies /mL at Week 60 | 0.993 | 0.988
  Proportion with VL<400 copies /mL at Week 72 | 0.996 | 0.988
  Proportion with VL<400 copies /mL at Week 84 | 0.988 | 0.994
  Proportion with VL<400 copies /mL at Week 96 | 1.000 | 0.987
  Proportion with VL<400 copies /mL at Week 108 | 0.996 | 1.000
  Proportion with VL<400 copies /mL at Week 120 | 1.000 | 0.994
  Proportion with VL<400 copies /mL at Week 132 | 0.996 | 0.993
  Proportion with VL<400 copies /mL at Week 144/EOT | 0.991 | 0.986

5. Secondary Outcome: Change in CD4+ Count From Baseline
Description: Change in CD4+ cell count from baseline among patients on treatment at each visit, with the final visit at Week 144 or EOT
Time Frame: From baseline to Weeks 4, 8, 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, 132 and 144/EOT
Population: FAS with varying numbers missing or not on treatment per visit
Measure: Mean (Standard Deviation); unit: cells/mm^3
Arm/Group | Nevirapine QD+BID | Atazanvir/Ritonavir
Number analyzed (Participants) | 376 | 193
cells/mm^3
  Change in CD4+ count to Week 4 | 77.2 (93.5) | 86.1 (94.4)
  Change in CD4+ count to Week 8 | 105.6 (108.0) | 98.0 (91.1)
  Change in CD4+ count to Week 12 | 120.3 (113.9) | 110.9 (111.6)
  Change in CD4+ count to Week 24 | 134.4 (114.9) | 133.8 (110.7)
  Change in CD4+ count to Week 36 | 160.1 (123.0) | 163.4 (119.8)
  Change in CD4+ count to Week 48 | 168.2 (127.0) | 183.6 (121.6)
  Change in CD4+ count to Week 60 | 184.8 (129.6) | 208.2 (144.2)
  Change in CD4+ count to Week 72 | 213.7 (165.7) | 231.9 (165.4)
  Change in CD4+ count to Week 84 | 223.0 (147.1) | 246.4 (149.4)
  Change in CD4+ count to Week 96 | 217.7 (133.5) | 251.6 (149.8)
  Change in CD4+ count to Week 108 | 231.2 (148.9) | 267.2 (161.2)
  Change in CD4+ count to Week 120 | 231.3 (147.6) | 269.2 (169.9)
  Change in CD4+ count to Week 132 | 243.4 (164.8) | 281.3 (147.3)
  Change in CD4+ count to Week 144/EOT | 251.0 (151.6) | 285.8 (164.8)

6. Secondary Outcome: Change in Framingham Score From Baseline
Description: Change in the estimated risk of cardiovascular disease using the Framingham algorithm from baseline to after 48, 96 and 144 weeks, last observation carried forward (LOCF). The score is based on age, gender, systolic blood pressure, total cholesterol, high density lipoprotein cholesterol and smoking status. Scores range from 0 to 21 with higher scores indicating a greater risk.
Time Frame: From baseline to Weeks 48, 96 and 144/EOT
Population: FAS with varying numbers missing
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Nevirapine QD+BID | Atazanvir/Ritonavir
Number analyzed (Participants) | 376 | 193
Units on a scale
  Change in Framingham score to Week 48 | 0.50 (2.79) | 0.66 (2.92)
  Change in Framingham score to Week 96 | 0.93 (3.15) | 1.19 (3.25)
  Change in Framingham score to Week 144/EOT | 1.14 (3.40) | 0.82 (3.03)

7. Secondary Outcome: Change in Mental Health Summary (MHS) Score From Baseline
Description: Quality of life (QoL) assessment by change in MHS score from baseline to after 48, 96 and 144 weeks (observed cases), from the Medical Outcomes Study HIV Health Survey (MOS-HIV), a 35-item self-administered questionnaire including 10 scales covering: health perceptions, pain, physical functioning, role functioning, social and cognitive functioning, mental health, energy/fatigue, health distress, and QoL. The MHS is a weighted average of the 10 scales and ranges from 0 to 100 with higher scores indicating better QoL.
Time Frame: From baseline to Weeks 48, 96 and 144/EOT
Population: FAS with varying numbers missing
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Nevirapine QD+BID | Atazanvir/Ritonavir
Number analyzed (Participants) | 376 | 193
Units on a scale
  Change in MHS score to Week 48 | 6.09 (9.31) | 4.52 (7.84)
  Change in MHS score to Week 96 | 6.10 (9.75) | 4.89 (9.58)
  Change in MHS score to Week 144/EOT | 4.76 (10.33) | 4.70 (10.14)

8. Secondary Outcome: Change in Physical Health Summary (PHS) Score From Baseline
Description: QoL assessment by change in PHS score from baseline to after 48, 96 and 144 weeks (observed cases), from the MOS-HIV, a 35-item self-administered questionnaire including 10 scales covering: health perceptions, pain, physical functioning, role functioning, social and cognitive functioning, mental health, energy/fatigue, health distress, and QoL. The PHS is a weighted average of the 10 scales and ranges from 0 to 100 with higher scores indicating better QoL.
Time Frame: From baseline to Weeks 48, 96 and 144/EOT
Population: FAS with varying numbers missing
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Nevirapine QD+BID | Atazanvir/Ritonavir
Number analyzed (Participants) | 376 | 193
Units on a scale
  Change in PHS score to Week 48 | 3.34 (7.77) | 3.35 (8.52)
  Change in PHS score to Week 96 | 3.19 (7.83) | 3.00 (7.34)
  Change in PHS score to Week 144/EOT | 2.22 (8.77) | 3.35 (8.42)

9. Secondary Outcome: Number of Patients Hospitalized
Description: Cost effectiveness assessment by number of patients hospitalized
Time Frame: From baseline to Week 24, Week 24 to 48, Week 48 to 96, and Week 96 to 144/EOT
Population: FAS with varying numbers missing
Measure: Number; unit: Patients
Arm/Group | Nevirapine QD+BID | Atazanvir/Ritonavir
Number analyzed (Participants) | 376 | 193
Patients
  Number hospitalized between baseline and Week 24 | 8 | 2
  Number hospitalized between Week 24 and Week 48 | 6 | 5
  Number hospitalized between Week 48 and Week 96 | 5 | 5
  Number hospitalized between Week 96 and Wk 144/EOT | 9 | 1

10. Secondary Outcome: Non-scheduled Physician Visits
Description: Cost effectiveness assessment by number of patients with non-scheduled physician visits
Time Frame: From baseline to Week 24, Week 24 to 48, Week 48 to 96, and Week 96 to 144/EOT
Population: FAS with varying numbers missing
Measure: Number; unit: patients
Arm/Group | Nevirapine QD+BID | Atazanvir/Ritonavir
Number analyzed (Participants) | 376 | 193
patients
  Number between baseline and Week 24 | 74 | 35
  Number between Week 24 and Week 48 | 45 | 35
  Number between Week 48 and Week 96 | 58 | 28
  Number between Week 96 and Wk 144/EOT | 58 | 35

11. Secondary Outcome: Genotypic Resistance Associated With Virologic Failure
Description: Number of treatment-emergent drug-associated substitutions in patients with virological failure up to Week 48. The total number of genotypic mutations in those patients who were virologic failures is given, not the number of patients with mutations.
Time Frame: From baseline to Week 48
Population: All patients with virologic failure assessed for genotypic resistance
Measure: Number; unit: Number of substitutions
Arm/Group | Nevirapine QD+BID | Atazanvir/Ritonavir
Number analyzed (Participants) | 30 | 2
Number of substitutions
  Emtricitabine-associated substitutions at Week 48 | 21 | 0
  Tenofovir-associated substitutions at Week 48 | 11 | 0
  Nevirapine-associated substitutions at Week 48 | 34 | 0

12. Secondary Outcome: Treatment-emergent AIDS-defining Illness
Description: Treatment-emergent AIDS-defining illness (tr.-emerg. AIDS-def.illness) including worsening during treatment
Time Frame: From baseline to Week 144
Population: FAS
Measure: Number; unit: Patients
Arm/Group | Nevirapine QD+BID | Atazanvir/Ritonavir
Number analyzed (Participants) | 376 | 193
Patients
  Number with tr.-emerg. AIDS-def.illness | 26 | 7
  Number without tr.-emerg. AIDS-def.illness | 350 | 186

13. Secondary Outcome: Treatment-emergent AIDS-defining Illness Leading to Death
Description: Patients with an AIDS-defining illness leading to death broken out by treatment. Statistical analysis shows time to death from AIDS-defining illness.
Time Frame: From baseline to Week 144
Population: FAS
Measure: Number; unit: Patients
Arm/Group | Nevirapine QD+BID | Atazanvir/Ritonavir
Number analyzed (Participants) | 376 | 193
Patients
  Number with AIDS-def. illness leading to death | 3 | 0
  Number without AIDS-def. illness leading to death | 373 | 193
Statistical Analysis 1: Comparison: Nevirapine QD+BID vs Atazanvir/Ritonavir; Test type: Superiority or Other; p = 0.0403, Regression, Cox; Hazard Ratio (HR) = 0.461, 95% CI [0.220 to 0.966]

14. Secondary Outcome: Lipodystrophy
Description: Number of patients with AE lipodystrophy
Time Frame: From baseline to Week 144
Population: FAS
Measure: Number; unit: Patients
Arm/Group | Nevirapine QD+BID | Atazanvir/Ritonavir
Number analyzed (Participants) | 376 | 193
Patients
  Number with lipodystrophy | 1 | 1
  Number without lipodystrophy | 375 | 192

15. Secondary Outcome: Serum Lipid Abnormalities
Description: Number of patients with AE elevated serum lipids (i.e. hypercholesterolaemia)
Time Frame: From baseline to Week 144
Population: FAS
Measure: Number; unit: patients
Arm/Group | Nevirapine QD+BID | Atazanvir/Ritonavir
Number analyzed (Participants) | 376 | 193
patients
  Number with serum lipid abnormalities | 9 | 4
  Number without serum lipid abnormalities | 367 | 189

16. Secondary Outcome: Glycaemic Abnormalities
Description: Number of patients with AE elevated serum glucose
Time Frame: From baseline to Week 144
Population: FAS
Measure: Number; unit: Patients
Arm/Group | Nevirapine QD+BID | Atazanvir/Ritonavir
Number analyzed (Participants) | 376 | 193
Patients
  Number with glycaemic abnormalities | 0 | 3
  Number without glycaemic abnormalities | 376 | 190

17. Secondary Outcome: Treatment Response at Week 96
Description: Treatment response is defined as a viral load (VL) <50 copies/mL measured at two consecutive visits prior to Week 96 and without subsequent rebound or change of antiretroviral (ARV) therapy prior to Week 96.
Time Frame: From baseline to Week 96
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Nevirapine QD | Nevirapine BID | Nevirapine QD+BID | Atazanvir/Ritonavir
Number analyzed (Participants) | 188 | 188 | 376 | 193
participants
  Number of responders | 131 | 122 | 253 | 149
  Number of non-responders | 57 | 66 | 123 | 44
Statistical Analysis 1: Comparison: Nevirapine QD+BID vs Atazanvir/Ritonavir; Test type: Non-Inferiority or Equivalence — Non-inferiority margin 12% (or 0.12 as proportion); p = 0.0109, Cochran-Mantel-Haenszel — Test for superiority following confirmation of non-inferiority; Analysis controlling for screening viral load and CD4+ count categories. N=373 NVP QD+BID patients and N=193 ATZ/r patients; Risk Difference (RD) = -0.097, 95% CI [-0.171 to -0.022]
Statistical Analysis 2: Comparison: Nevirapine QD vs Atazanvir/Ritonavir; Test type: Non-Inferiority or Equivalence — Non-inferiority margin 12% (or 0.12 as proportion); p = 0.1033, Cochran-Mantel-Haenszel — Test for superiority following confirmation of non-inferiority; Analysis controlling for screening viral load and CD4+ count categories. N=186 NVP QD patients and N=193 ATZ/r patients; Risk Difference (RD) = -0.072, 95% CI [-0.158 to 0.015]
Statistical Analysis 3: Comparison: Nevirapine BID vs Atazanvir/Ritonavir; Test type: Non-Inferiority or Equivalence — Non-inferiority margin 12% (or 0.12 as proportion); p = 0.0073, Cochran-Mantel-Haenszel — Test for superiority following confirmation of non-inferiority; Analysis controlling for screening viral load and CD4+ count categories. N=187 NVP QD patients and N=193 ATZ/r patients; Risk Difference (RD) = -0.122, 95% CI [-0.212 to -0.033]

18. Secondary Outcome: Treatment Response at Week 144
Description: Treatment response is defined as a viral load (VL) <50 copies/mL measured at two consecutive visits prior to Week 144 and without subsequent rebound or change of antiretroviral (ARV) therapy prior to Week 144.
Time Frame: From baseline to Week 144
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Nevirapine QD | Nevirapine BID | Nevirapine QD+BID | Atazanvir/Ritonavir
Number analyzed (Participants) | 188 | 188 | 376 | 193
participants
  Number of responders | 121 | 113 | 234 | 143
  Number of non-responders | 67 | 75 | 142 | 50
Statistical Analysis 1: Comparison: Nevirapine QD+BID vs Atazanvir/Ritonavir; Test type: Non-Inferiority or Equivalence — Non-inferiority margin 12% (or 0.12 as proportion); p = 0.0031, Cochran-Mantel-Haenszel — Test for superiority following confirmation of non-inferiority; [statistical method as in outcome 17, analysis 1]; Risk Difference (RD) = -0.117, 95% CI [-0.194 to -0.040]
Statistical Analysis 2: Comparison: Nevirapine QD vs Atazanvir/Ritonavir; Test type: Non-Inferiority or Equivalence — Non-inferiority margin 12% (or 0.12 as proportion); p = 0.0365, Cochran-Mantel-Haenszel — Test for superiority following confirmation of non-inferiority; Analysis controlling for screening viral load and CD4+ count categories. N=186 NVP QD patients and N=193 ATZ/r patients; Risk Difference (RD) = -0.096, 95% CI [-0.186 to -0.006]
Statistical Analysis 3: Comparison: Nevirapine BID vs Atazanvir/Ritonavir; Test type: Non-Inferiority or Equivalence — Non-inferiority margin 12% (or 0.12 as proportion); p = 0.0033, Cochran-Mantel-Haenszel — Test for superiority following confirmation of non-inferiority; Analysis controlling for screening viral load and CD4+ count categories. N=187 NVP QD patients and N=193 ATZ/r patients; Risk Difference (RD) = -0.139, 95% CI [-0.231 to -0.046]

19. Secondary Outcome: Proportion of Patients With Virological Rebound With VL >=50 Copies/mL After CVR (Confirmed Virological Response) at Week 24, 48, 96, 144
Description: The analyses of virologic rebound were performed on the original values at each visit(ORGV) rather than calculated results within time windows (CAL)
Time Frame: at Week 24, 48, 96, 144
Population: Full Analysis Set (FAS) defined as all randomized and treated patients.
Measure: Number; unit: participants
Arm/Group | Nevirapine QD | Nevirapine BID | Nevirapine QD+BID | Atazanvir/Ritonavir
Number analyzed (Participants) | 188 | 188 | 376 | 193
participants
  virologic rebound after CVR at Week 24 | 3 | 2 | 5 | 5
  virologic rebound after CVR at Week 48 | 4 | 5 | 9 | 12
  virologic rebound after CVR at Week 96 | 4 | 6 | 10 | 10
  virologic rebound after CVR at Week 144 | 8 | 9 | 17 | 15

20. Secondary Outcome: Proportion of Patients With Virological Rebound With VL >=400 Copies/mL After CVR at Week 24, 48, 96, 144
Description: as for outcome 19
Time Frame: at Week 24, 48, 96, 144
Population: Full Analysis Set (FAS) defined as all randomized and treated patients.
Measure: Number; unit: participants
Arm/Group | Nevirapine QD | Nevirapine BID | Nevirapine QD+BID | Atazanvir/Ritonavir
Number analyzed (Participants) | 188 | 188 | 376 | 193
participants
  virologic rebound after CVR at Week 24 | 2 | 2 | 4 | 2
  virologic rebound after CVR at Week 48 | 3 | 3 | 6 | 2
  virologic rebound after CVR at Week 96 | 3 | 6 | 9 | 2
  virologic rebound after CVR at Week 144 | 4 | 6 | 10 | 5

21. Secondary Outcome: Proportion of Patients With Virologic Failure at Week 48, 96, 144
Time Frame: at Week 48, 96, 144
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Nevirapine QD | Nevirapine BID | Nevirapine QD+BID | Atazanvir/Ritonavir
Number analyzed (Participants) | 188 | 188 | 376 | 193
participants
  virologic failure at Week 48 | 20 | 25 | 45 | 25
  virologic failure at Week 96 | 15 | 25 | 40 | 13
  virologic failure at Week 144 | 19 | 28 | 47 | 17
Statistical Analysis 1: Comparison: Nevirapine BID vs Atazanvir/Ritonavir; week 48; Test type: Non-Inferiority or Equivalence — H0: Difference in proportions = 0; p = 0.9784, Cochran Chi-Squared; Difference in proportions = 0.001, 95% CI 2-sided [-0.065 to 0.066]
Statistical Analysis 2: Comparison: Nevirapine BID vs Atazanvir/Ritonavir; week 96; Test type: Non-Inferiority or Equivalence — H0: Difference in proportions = 0; p = 0.0331, Cochran Chi-Squared; Difference in proportions = 0.064, 95% CI 2-sided [0.005 to 0.123]
Statistical Analysis 3: Comparison: Nevirapine BID vs Atazanvir/Ritonavir; week 144; Test type: Non-Inferiority or Equivalence — H0: Difference in proportions = 0; p = 0.0691, Cochran Chi-Squared; Difference in proportions = 0.058, 95% CI 2-sided [-0.005 to 0.121]
Statistical Analysis 4: Comparison: Nevirapine QD vs Atazanvir/Ritonavir; week 48; Test type: Non-Inferiority or Equivalence — H0: Difference in proportions = 0; p = 0.4585, Cochran Chi-Squared; Difference in proportions = -0.023, 95% CI 2-sided [-0.084 to 0.038]
Statistical Analysis 5: Comparison: Nevirapine QD vs Atazanvir/Ritonavir; week 96; Test type: Non-Inferiority or Equivalence — H0: Difference in proportions = 0; p = 0.5438, Cochran Chi-Squared; Difference in proportions = 0.015, 95% CI 2-sided [-0.034 to 0.064]
Statistical Analysis 6: Comparison: Nevirapine QD vs Atazanvir/Ritonavir; week 144; Test type: Non-Inferiority or Equivalence — H0: Difference in proportions = 0; p = 0.5659, Cochran Chi-Squared; Difference in proportions = 0.016, 95% CI 2-sided [-0.039 to 0.071]

22. Secondary Outcome: Time to Treatment Response (First Confirmed VL<50 Copies/mL)
Description: Time to treatment response was defined as the time from start of treatment until the first measurement of the first confirmed virological response
Time Frame: baseline to week 144
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: weeks
Arm/Group | Nevirapine QD | Nevirapine BID | Nevirapine QD+BID | Atazanvir/Ritonavir
Number analyzed (Participants) | 188 | 188 | 376 | 193
weeks | 12.00 [8.00 to 24.00] | 12.14 [8.00 to 24.00] | 12.00 [8.00 to 24.00] | 23.71 [11.29 to 25.14]
Statistical Analysis 1: Comparison: Nevirapine QD+BID vs Atazanvir/Ritonavir; Test type: Superiority or Other; p = 0.0002, Regression, Cox; Hazard Ratio (HR) = 0.692, 95% CI [0.570 to 0.839]
Statistical Analysis 2: Comparison: Nevirapine QD+BID vs Atazanvir/Ritonavir; Cox regression on responders only (N=289 in Nevirapine QD+BID and N=175 in Atazanvir/ritonavir); Test type: Superiority or Other; p < 0.0001, Regression, Cox; Hazard Ratio (HR) = 0.630, 95% CI [0.519 to 0.764]

23. Secondary Outcome: Time to Loss of Virologic Response (Rebound)
Description: Time to loss of virologic response (TLOVR) was defined as the time from start of treatment to the first measurement showing VL ≥ 50 copies/mL in the first virologic rebound, after having a confirmed virological response.
Time Frame: Baseline to week 144
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: weeks
Arm/Group | Nevirapine QD | Nevirapine BID | Nevirapine QD+BID | Atazanvir/Ritonavir
Number analyzed (Participants) | 188 | 188 | 376 | 193
weeks | 143.86 [48.43 to 144.00] | 143.21 [0.00 to 144.00] | 143.71 [4.29 to 144.00] | 143.00 [119.29 to 144.00]
Statistical Analysis 1: Comparison: Nevirapine QD+BID vs Atazanvir/Ritonavir; Test type: Superiority or Other; p = 0.1329, Regression, Cox; Hazard Ratio (HR) = 0.762, 95% CI [0.535 to 1.086]

24. Secondary Outcome: Time to Treatment Failure
Description: Treatment failure is defined as the occurrence of the first of at least one of the following events: early discontinuation of trial drug, change in ARV therapy, failure to achieve an HIV RNA count < 50 copies/mL up to Visit 10 (week 48) or loss of virologic response
Time Frame: baseline to week 144
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: weeks
Arm/Group | Nevirapine QD | Nevirapine BID | Nevirapine QD+BID | Atazanvir/Ritonavir
Number analyzed (Participants) | 188 | 188 | 376 | 193
weeks | 143.86 [48.43 to 144.00] | 143.21 [0.00 to 144.00] | 143.71 [30.07 to 144.00] | 143.00 [119.29 to 144.00]
Statistical Analysis 1: Comparison: Nevirapine QD+BID vs Atazanvir/Ritonavir; Test type: Superiority or Other; p = 0.0444, Regression, Cox; Hazard Ratio (HR) = 0.731, 95% CI [0.539 to 0.992]

25. Secondary Outcome: Change in the Calculated Glomerular Filtration Rate (GFR) at Week 48, 96 and 144
Description: Calculations based on the MDRD algorithm.
Time Frame: From baseline to Week 48, 96, 144
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mL/min/1.73 m^2
Arm/Group | Nevirapine QD | Nevirapine BID | Nevirapine QD+BID | Atazanvir/Ritonavir
Number analyzed (Participants) | 188 | 188 | 376 | 193
mL/min/1.73 m^2
  change baseline to week 48 (N=143, 128, 271, 173) | -3.91 (13.93) | -5.92 (17.11) | -4.86 (15.52) | -7.18 (15.19)
  change baseline to week 96 (N=130, 122, 252, 157) | -6.93 (14.33) | -10.02 (17.37) | -8.42 (15.92) | -11.53 (15.59)
  change baseline to week 144 (N=163, 168, 331, 174) | -3.27 (20.65) | -6.33 (17.30) | -4.82 (19.06) | -9.56 (17.47)

26. Secondary Outcome: Proportion of Patients With >= DAIDS Grade 2 Laboratory Abnormalities
Time Frame: week 148
Population: Full Analysis Set (FAS) defined as all randomized and treated patients.
Measure: Number; unit: participants
Groups:
- Nevirapine QD: NVP 400mg QD on a background of the fixed combination Truvada®
Arm/Group | Nevirapine QD | Nevirapine BID | Atazanvir/Ritonavir
Number analyzed (Participants) | 188 | 188 | 193
participants
  DAIDS 2 moderate | 74 | 84 | 72
  DAIDS 3 severe | 30 | 28 | 39
  DAIDS 4 potential lifethreatening | 9 | 15 | 9

27. Secondary Outcome: Proportion of Patients Reporting Rash of Any Severity
Description: Proportion of Patients reporting rash of any severity
Time Frame: week 148
Population: Full Analysis Set (FAS) defined as all randomized and treated patients.
Measure: Number; unit: participants
Arm/Group | Nevirapine QD | Nevirapine BID | Atazanvir/Ritonavir
Number analyzed (Participants) | 188 | 188 | 193
participants | 75 | 64 | 74

28. Secondary Outcome: Proportion of Patients Reporting Hepatic Events of Any Severity
Description: Proportion of Patients reporting hepatic events of any severity
Time Frame: week 148
Population: Full Analysis Set (FAS) defined as all randomized and treated patients.
Measure: Number; unit: participants
Arm/Group | Nevirapine QD | Nevirapine BID | Atazanvir/Ritonavir
Number analyzed (Participants) | 188 | 188 | 193
participants | 26 | 24 | 92

29. Secondary Outcome: Proportion of Patients Reporting CNS (Central Nervous System) Side Effects of Any Severity
Description: Proportion of Patients reporting CNS (central nervous system) side effects of any severity
Time Frame: week 148
Population: Full Analysis Set (FAS) defined as all randomized and treated patients.
Measure: Number; unit: participants
Arm/Group | Nevirapine QD | Nevirapine BID | Atazanvir/Ritonavir
Number analyzed (Participants) | 188 | 188 | 193
participants | 41 | 41 | 37

30. Secondary Outcome: Change of Cholesterol Values From Baseline to Week 48, 96, 144
Description: Changes frombaseline in total cholesterol, LDL-cholesterol(LDL-c) and HDL
Time Frame: baseline to week 48, 96, 144
Population: FAS, where only patients with corresponding laboratory values for the considered time point are considered
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Nevirapine QD | Nevirapine BID | Atazanvir/Ritonavir
Number analyzed (Participants) | 188 | 188 | 193
mg/dL
  total cholesterol, week 48 (N=138,122,164) | 29.28 (30.64) | 29.54 (27.33) | 20.84 (30.46)
  total cholesterol, week 96 (N=124,114,147) | 39.17 (33.67) | 36.87 (30.60) | 29.99 (31.93)
  total cholesterol, week 144 (N=154,155,160) | 33.12 (32.77) | 30.66 (33.24) | 28.13 (32.06)
  LDL-c, week 48 (N=136,117,159) | 16.54 (24.44) | 17.70 (22.16) | 10.58 (26.07)
  LDL-c, week 96 (N=119,110,145) | 21.93 (23.44) | 21.66 (25.14) | 19.19 (25.49)
  LDL-c, week 144 (N=151,150,157) | 21.42 (26.61) | 17.95 (26.04) | 17.61 (28.33)
  HDL, week 48(N=138,122,164) | 12.06 (9.72) | 11.59 (10.95) | 3.49 (9.44)
  HDL, week 96 (N=124,114,147) | 13.86 (10.95) | 13.33 (12.00) | 4.74 (10.62)
  HDL, week 144(N=154,155,160) | 12.61 (13.64) | 10.47 (15.35) | 5.73 (11.14)

31. Secondary Outcome: Changes of Apolipoprotein Values From Baseline to Week 48, 96, 144
Description: Changes frombaseline apolipoprotein A1 & B
Time Frame: baseline to week 48, 96, 144
Population: FAS, where only patients with corresponding laboratory values for the considered time point are considered
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Nevirapine QD | Nevirapine BID | Atazanvir/Ritonavir
Number analyzed (Participants) | 188 | 188 | 193
g/L
  apolipoprotein A1, week 48 (N=134,121,156) | 0.23 (0.22) | 0.23 (0.24) | 0.08 (0.21)
  apolipoprotein A1, week 96 (N=115,106,141) | 0.23 (0.24) | 0.23 (0.25) | 0.07 (0.22)
  apolipoprotein A1, week 144 (N=144,140,148) | 0.16 (0.24) | 0.14 (0.26) | 0.06 (0.23)
  apolipoprotein B, week 48 (N=134,120,156) | 0.00 (0.17) | 0.03 (0.16) | 0.03 (0.16)
  apolipoprotein B, week 96 (N=115,106,141) | 0.00 (0.16) | -0.00 (0.17) | 0.03 (0.17)
  apolipoprotein B, week 144 (N=144,139,148) | 0.01 (0.16) | 0.05 (0.18) | 0.03 (0.17)

32. Secondary Outcome: Change of hsCRP From Baseline to Week 48, 96, 144
Description: Change of hsCRP from baseline to week 48, 96, 144
Time Frame: baseline to week 48, 96, 144
Population: FAS, where only patients with corresponding laboratory values for the considered time point are considered
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Nevirapine QD | Nevirapine BID | Atazanvir/Ritonavir
Number analyzed (Participants) | 188 | 188 | 193
mg/L
  hsCRP, week 48 (N=142,126,173) | -1.01 (12.53) | -0.67 (12.71) | -0.70 (8.61)
  hsCRP, week 96 (N=128,120,157) | -1.54 (11.21) | -0.79 (21.32) | 0.35 (15.19)
  hsCRP, week 144 (N=160,164,174) | -0.09 (14.34) | -0.02 (12.76) | 0.04 (8.20)

33. Secondary Outcome: Change of Total Triglycerides From Baseline to Week 48, 96, 144
Description: Change of total triglycerides from baseline to week 48, 96, 144
Time Frame: baseline to week 48, 96, 144
Population: FAS, where only patients with corresponding laboratory values for the considered time point are considered
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Nevirapine QD | Nevirapine BID | Atazanvir/Ritonavir
Number analyzed (Participants) | 188 | 188 | 193
mg/dL
  total triglycerides, week 48 (N=138,120,164) | 0.08 (92.39) | 1.67 (99.31) | 36.28 (80.24)
  total triglycerides, week 96 (N=124,113,147) | 9.34 (95.66) | 5.35 (84.92) | 30.45 (94.99)
  total triglycerides, week 144 (N=153,153,159) | -3.46 (77.97) | 6.11 (80.82) | 27.11 (85.97)

34. Secondary Outcome: Change of Total Cholesterol to HDL-cholesterol Ratio From Baseline to Week 48, 96, 144
Description: Change of Total cholesterol to HDL-cholesterol ratio from baseline to week 48, 96, 144
Time Frame: baseline to week 48, 96, 144
Population: FAS, where only patients with corresponding laboratory values for the considered time point are considered
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Nevirapine QD | Nevirapine BID | Atazanvir/Ritonavir
Number analyzed (Participants) | 188 | 188 | 193
ratio
  total triglycerides, week 48 (N=138,122,164) | -0.37 (0.95) | -0.33 (1.05) | 0.20 (0.99)
  total triglycerides, week 96 (N=124,114,147) | -0.22 (0.93) | -0.25 (1.03) | 0.28 (1.05)
  total triglycerides, week 144 (N=154,155,160) | -0.24 (0.96) | -0.07 (1.45) | 0.17 (1.05)

ADVERSE EVENTS:
Time Frame: 148 weeks
Arm/Group | Nevirapine QD | Nevirapine BID | Atazanvir/Ritonavir
Serious Adverse Events (participants affected / at risk) | 25/188 | 31/188 | 27/193
Other Adverse Events (participants affected / at risk) | 136/188 | 141/188 | 161/193
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nevirapine QD (N=188) | Nevirapine BID (N=188) | Atazanvir/Ritonavir (N=193)
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 1 | 0
Angina unstable (Cardiac disorders) | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1
Myopericarditis (Cardiac disorders) | 0 | 1 | 0
Goitre (Endocrine disorders) | 1 | 0 | 0
Retinal detachment (Eye disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0
Peritonitis (Gastrointestinal disorders) | 0 | 1 | 0
Asthenia (General disorders) | 0 | 1 | 0
Fatigue (General disorders) | 0 | 1 | 0
Multi-organ failure (General disorders) | 1 | 0 | 0
Pain (General disorders) | 0 | 1 | 0
Puncture site haemorrhage (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 3 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 3 | 0
Cholestasis (Hepatobiliary disorders) | 1 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0 | 0
Abscess jaw (Infections and infestations) | 1 | 0 | 0
Anal abscess (Infections and infestations) | 1 | 0 | 0
Anogenital warts (Infections and infestations) | 0 | 0 | 5
Appendicitis (Infections and infestations) | 0 | 1 | 0
Candida pneumonia (Infections and infestations) | 0 | 1 | 0
Cerebral toxoplasmosis (Infections and infestations) | 1 | 0 | 0
Cryptococcosis (Infections and infestations) | 1 | 0 | 0
Cytomegalovirus infection (Infections and infestations) | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 1
H1N1 influenza (Infections and infestations) | 1 | 0 | 0
HIV infection (Infections and infestations) | 0 | 1 | 0
Hepatitis A (Infections and infestations) | 0 | 0 | 2
Herpes zoster (Infections and infestations) | 1 | 0 | 0
Meningitis viral (Infections and infestations) | 0 | 0 | 1
Neurosyphilis (Infections and infestations) | 1 | 0 | 0
Orchitis (Infections and infestations) | 0 | 0 | 1
Papilloma viral infection (Infections and infestations) | 0 | 1 | 0
Pneumocystis jiroveci pneumonia (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 0 | 3
Postoperative wound infection (Infections and infestations) | 1 | 0 | 0
Pulmonary tuberculosis (Infections and infestations) | 1 | 0 | 0
Salpingitis (Infections and infestations) | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 1
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 1
Tuberculosis (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1
Drug exposure during pregnancy (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 1 | 0
Fracture of penis (Injury, poisoning and procedural complications) | 0 | 0 | 1
Meniscus lesion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Multiple injuries (Injury, poisoning and procedural complications) | 0 | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 2 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 1 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 0
Haemoglobin decreased (Investigations) | 1 | 0 | 0
Transaminases increased (Investigations) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Bone neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2 | 0
Kaposi's sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Lung carcinoma cell type unspecified recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Carpal tunnel syndrome (Nervous system disorders) | 1 | 0 | 0
Cerebellar syndrome (Nervous system disorders) | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 2 | 0
Convulsion (Nervous system disorders) | 0 | 1 | 0
Epilepsy (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0
Neuralgia (Nervous system disorders) | 1 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 1 | 0
Alcohol abuse (Psychiatric disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0
Schizophrenia (Psychiatric disorders) | 0 | 1 | 0
Suicide attempt (Psychiatric disorders) | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 1 | 0
Cervical dysplasia (Reproductive system and breast disorders) | 1 | 0 | 0
Ovarian cyst ruptured (Reproductive system and breast disorders) | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Breast prosthesis implantation (Surgical and medical procedures) | 0 | 1 | 0
Mastoidectomy (Surgical and medical procedures) | 0 | 0 | 1
Tympanoplasty (Surgical and medical procedures) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nevirapine QD (N=188) | Nevirapine BID (N=188) | Atazanvir/Ritonavir (N=193)
Ocular icterus (Eye disorders) | 0 | 0 | 14
Abdominal pain (Gastrointestinal disorders) | 5 | 10 | 15
Abdominal pain upper (Gastrointestinal disorders) | 9 | 14 | 13
Diarrhoea (Gastrointestinal disorders) | 29 | 33 | 47
Flatulence (Gastrointestinal disorders) | 9 | 10 | 9
Nausea (Gastrointestinal disorders) | 22 | 21 | 21
Vomiting (Gastrointestinal disorders) | 13 | 15 | 8
Fatigue (General disorders) | 11 | 11 | 12
Influenza like illness (General disorders) | 10 | 6 | 9
Pyrexia (General disorders) | 14 | 13 | 9
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 15
Jaundice (Hepatobiliary disorders) | 0 | 0 | 40
Bronchitis (Infections and infestations) | 28 | 19 | 19
Gastroenteritis (Infections and infestations) | 8 | 14 | 8
Gonorrhoea (Infections and infestations) | 11 | 3 | 4
Herpes zoster (Infections and infestations) | 16 | 12 | 7
Influenza (Infections and infestations) | 21 | 18 | 16
Nasopharyngitis (Infections and infestations) | 41 | 36 | 40
Pharyngitis (Infections and infestations) | 10 | 10 | 12
Rhinitis (Infections and infestations) | 8 | 7 | 13
Sinusitis (Infections and infestations) | 13 | 9 | 10
Upper respiratory tract infection (Infections and infestations) | 6 | 8 | 14
Blood bilirubin increased (Investigations) | 0 | 1 | 33
Arthralgia (Musculoskeletal and connective tissue disorders) | 14 | 8 | 11
Back pain (Musculoskeletal and connective tissue disorders) | 14 | 13 | 17
Myalgia (Musculoskeletal and connective tissue disorders) | 12 | 10 | 9
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 11
Headache (Nervous system disorders) | 27 | 24 | 35
Depression (Psychiatric disorders) | 16 | 9 | 18
Cough (Respiratory, thoracic and mediastinal disorders) | 18 | 22 | 21
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 | 4 | 12
Rash (Skin and subcutaneous tissue disorders) | 25 | 31 | 23
Hypertension (Vascular disorders) | 10 | 9 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Other - Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.